CLINICAL TRIAL: NCT01166646
Title: Blinded Study of Topical Investigational Lotion Vs. Approved Cream in Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000-0551-202
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — halobetasol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Halobetasol Proprionate Lotion 0.05% (Experimental): Subjects randomized to receive lotion
  Interventions: Drug: Halobetasol Proprionate Lotion 0.05%
- Halobetasol Proprionate Cream 0.05% (Active Comparator): Subjects randomized to receive cream
  Interventions: Drug: Halobetasol Proprionate Cream 0.05%

INTERVENTIONS:
Drug: Halobetasol Proprionate Lotion 0.05% — Apply 3.5 grams twice daily for 1-2 weeks
  Arms: Halobetasol Proprionate Lotion 0.05%
Drug: Halobetasol Proprionate Cream 0.05% — Apply 3.5 grams twice daily for 1-2 weeks
  Other Names: Ultravate
  Arms: Halobetasol Proprionate Cream 0.05%

SUMMARY:
The purpose of this study is to determine whether the investigational lotion is an effective treatment of moderate to severe plaque psoriasis in comparison to an approved cream.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are male or non-pregnant female; 18 years of age at the time of screening.
* Subjects provide Institutional Review Board (IRB) approved written informed consent for participating in this study.
* Subjects have a clinical diagnosis of stable plaque psoriasis involving a minimum of 20% body surface area and an Overall Disease Severity (ODS) score on the designated treatment area of at least 3 as determined by the evaluating investigator.
* Subjects are willing and able to apply the study medication as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at the Screening (Part B) and Baseline Visits and agree to use an effective form of birth control for the duration of the study (abstinence, stabilized on oral contraceptives or contraceptive patches for at least three months, implant, injection, IUD, NuvaRing®, condom and spermicidal or diaphragm and spermicidal). Abstinence is an acceptable form of birth control for subjects who are not sexually active. Subjects who become sexually active during the trial must agree to use an effective, non-prohibited form of birth control for the duration of the study.

Exclusion Criteria:

* Subjects have spontaneously improving or rapidly deteriorating plaque psoriasis, or have guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
* Subjects have a physical condition which, in the Investigator's opinion, might impair evaluation of plaque psoriasis, adrenal axis function (e.g., Addison's Disease, Cushing's Syndrome) or which exposes the subject to an unacceptable risk by study participation.
* Subjects have used any phototherapy (including laser), photo-chemotherapy or systemic psoriasis therapy including methotrexate, retinoids, cyclosporine or biologics within 30 days prior to the initiation of study medication treatment.
* Subjects have used systemic corticosteroids (including oral or intramuscular) or topical, inhaled or intranasal corticosteroids within 30 or 14 days, respectively, prior to Part B of the Screening Visit and/or subjects have used systemic or topical corticosteroids between the Screening Visit and the initiation of treatment.
* Subjects have had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the initiation of treatment or are intending to have such exposure during the study that is thought by the Investigator to likely modify the subject's disease.
* Subjects have used topical psoriatic therapy including tar, anthralin, retinoids, vitamin D analogs (e.g., Dovonex®) within 14 days prior to the initiation of study medication treatment.
* Subjects have used emollients/moisturizers on areas to be treated within one day prior to the initiation of study medication treatment.
* Subjects are currently using lithium or plaquenil.
* Subjects are currently using a beta-blocking medication (e.g., propanolol) or angiotensin converting enzyme (ACE) inhibitors at a dose that has not been stabilized, in the opinion of the Investigator.
* Subjects have a history of sensitivity to any of the ingredients in the study medication.
* Subjects are pregnant, nursing or planning a pregnancy during the study period.
* Subjects are currently enrolled in an investigational drug or device study.
* Subjects have received an investigational drug or an investigational device within 30 days prior to screening.
* Subjects have been previously enrolled in this study and treated with the study medication.
* Subjects have irregular sleep schedules or work night shifts (cortisol levels exhibit physiological diurnal variation).
* Subjects have a screening CST with a post 30-minute stimulation cortisol level of ≤ 18 µg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Therapeutics Clinical Research, San Diego, California
  - Michigan Center for Skin Care Research (dba Skin Care Research), Clinton Township, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Dermatology, Laser & Vein Specialists of the Carolinas PLLC, Charlotte, North Carolina
  - DermResearch Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 2010 to May 2011
  The location of clinical sites included private dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Groups:
- Halobetasol Proprionate Lotion 0.05%: Subjects randomized to receive lotion
  Halobetasol Proprionate Lotion 0.05%: Apply 3.5 grams twice daily for up to 2 weeks
- Halobetasol Proprionate Cream 0.05%: Subjects randomized to receive cream
  Halobetasol Proprionate Cream 0.05%: Apply 3.5 grams twice daily for up to 2 weeks
Period: Overall Study
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Started | 21 | 22
Completed | 20 | 21
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) population included all participants enrolled in the study who were dispensed and applied test article at least once and had at least one follow-up visit after the Baseline visit (Visit 2). All 43 enrolled subjects were included in the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05% | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (9.28) | 47.7 (12.57) | 48.5 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 16 | 20 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adrenal Suppression Potential
Description: Hypothalamic Pituitary-Adrenal (HPA)-Axis responses to Cosyntropin Stimulation Testing (CST) were dichotomized to normal and abnormal. An abnormal HPA Axis response (HPA Suppression) was defined as a 30-minute post-stimulation serum cortisol level of ≤18 μg/dL at the end of treatment.
Time Frame: After 1-2 weeks dose
Population: Analysis shown is based on the ITT population, defined as all enrolled participants who were randomized and applied at least one dose of the test article.
Measure: Number; unit: participants
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 21 | 21
participants
  Normal | 16 | 18
  Abnormal | 5 | 3

2. Primary Outcome: Pharmacokinetic Properties (Cmax)
Description: Comparison of PK results (peak concentration in plasma [Cmax]) between the two Treatment Groups will be conducted following the last application of the medication on Day 8.
Time Frame: Day 8
Population: Pharmacokinetic properties were evaluated in a subgroup of 12 adult subjects per arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 12 | 12
pg/mL | 145.9 (106.9) | 136.2 (71.44)

3. Primary Outcome: Pharmacokinetic Properties (Tmax)
Description: Comparison of PK results (time to peak concentration [Tmax]) between the two Treatment Groups will be conducted following the last application of the medication on Day 8.
Time Frame: Day 8
Population: Pharmacokinetic properties were evaluated in a subgroup of 12 adult subjects per arm.
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 12 | 12
Hours | 3 [0 to 6] | 3 [0 to 8]

4. Primary Outcome: Pharmacokinetic Properties (AUC)
Description: Comparison of PK results (area under the curve [AUC] from time 0 to infinity) between the two Treatment Groups will be conducted following the last application of the medication on Day 8.
Time Frame: Day 8
Population: Pharmacokinetics properties were evaluated in a subgroup of 12 adult subjects per arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 12 | 12
pg*h/mL | 1267.7 (89.84) | 1229.8 (67.19)

5. Secondary Outcome: Changes in Disease Severity (Success)
Description: Overall disease severity (ODS) will be recorded at baseline, Day 8, and Day 15 on a 0 (clear) to 4 (severe/very severe) point scale. ODS evaluations will be dichotomized to "success" and "failure" with success defined as a grade of 1 or 0 at the end of treatment (EOT).
Time Frame: Day 15
Population: Analysis shown is based on the ITT population at Day 15.
Measure: Number; unit: participants
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 21 | 22
participants | 1 | 5

6. Secondary Outcome: Number of Subjects Whose Signs of Psoriasis Was Designated "Success"
Description: Signs of psoriasis including scaling, erythema, and plaque elevation will be recorded at baseline, Day 8, and Day 15 on a 0 (clear) to 4 (severe/very severe) point scale. Each of the signs of psoriasis will be dichotomized to a) "success" and "failure" with success defined as a grade of 1 or 0 at the End of Treatment (EOT; i.e., the visit at which psoriasis has cleared [Day 8 or Day 15] or end of the assigned treatment period).
Time Frame: Day 15
Population: Analysis shown is based on the number of subjects whose Signs of Psoriasis was designated "Success" (ITT population) at Day 15.
Measure: Number; unit: participants
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Number analyzed (Participants) | 21 | 22
participants
  Scaling | 6 | 11
  Erythema | 2 | 6
  Plaque elevation | 2 | 7

ADVERSE EVENTS:
Time Frame: AEs were collected from study screening (performed 14 days prior to baseline/first dose) to end of study treatment or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The Safety population included all subjects enrolled in the study who were dispensed the test article at least once.
Arm/Group | Halobetasol Proprionate Lotion 0.05% | Halobetasol Proprionate Cream 0.05%
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 9/21 | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Halobetasol Proprionate Lotion 0.05% (N=21) | Halobetasol Proprionate Cream 0.05% (N=22)
Type 2 diabetes mellitus (Endocrine disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Application site pain (General disorders) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Pallor (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Throat infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACTH stimulation test abnormal (Investigations) | 5 (5) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public dissemination. The PI may not disclose previously undisclosed confidential information other than study results.